CLINICAL TRIAL: NCT01479244
Title: PRESENT: Prevention of Recurrence in Early-Stage, Node-Positive Breast Cancer With Low to Intermediate HER2 Expressions With NeuVax™Treatment
Brief Title: Efficacy and Safety Study of NeuVax™ (Nelipepimut-S or E75) Vaccine to Prevent Breast Cancer Recurrence
Acronym: PRESENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galena Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NeuVax™ PH3-01, BB-IND 009187; 2011-005219-98 (EudraCT Number)
Record Dates: First submitted 2011-11-20; First posted 2011-11-24 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer With Low to Intermediate HER2 Expression
Keywords: HER2; low or intermediate; breast cancer; node-positive tumors
MeSH Terms: conditions — Breast Neoplasms | interventions — HER2 peptide (369-377); sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NeuVax™ (Experimental): NeuVax™ in WFI solution with Leukine®
  Interventions: Biological: NeuVax™ vaccine
- Leukine® (Active Comparator): Leukine® with WFI
  Interventions: Biological: Leukine® (sargramostim, GM-CSF) and water for injection

INTERVENTIONS:
Biological: NeuVax™ vaccine — E75 peptide acetate (HER2/neu p366-379) in WFI (1.5 mg/mL) mixed with 250 micrograms Leukine® (sargramostim, GM-CSF), will be administered in intradermal injections, in four divided doses (4 sites on upper thigh) once a month, for six consecutive months. At the end of the six months, NeuVax™ vaccine boosters will be given the same way once every six months for the next five times (totaling 36 months).
  Other Names: E75 peptide acetate , WFI, sargramostim, GM-CSF
  Arms: NeuVax™
Biological: Leukine® (sargramostim, GM-CSF) and water for injection — Leukine® 250 micrograms in water for injection, will be administered in intradermal injections, in four divided doses (4 sites on upper thigh) once a month, for six consecutive months. At the end of the six months, boosters inoculations will be given the same way once every six months for the next five times (totaling 36 months).
  Other Names: Leukine®
  Arms: Leukine®

SUMMARY:
Purpose of this trial:

1. To assess the efficacy and safety of NeuVax™ administered with adjuvant Leukine® (sargramostim, GM-CSF).
2. To evaluate and compare the disease free survival (DFS) in the vaccinated and control subjects.

DETAILED DESCRIPTION:
This is a multicenter, multinational, prospective, randomized, double-blind, controlled Phase 3 study.

The subjects eligible for this trial have an early stage node-positive breast cancer. Their tumors express low or intermediate levels of the HER2 protein. NeuVax™ will be administered after completion of front-line, standard of care therapy (surgery, radiation therapy, and chemotherapy) and can be given concomitantly with physician prescribed endocrine treatment.

NeuVax™ is the immmunodominant nonapeptide derived from the extracellular domain of the HER2 protein, a well-established target for therapeutic intervention in breast carcinoma. The nelipepimut sequence stimulates specific CD8+ cytotoxic T lymphocytes (CTL) following binding to HLA-A2/A3 molecules on antigen presenting cells (APC). These activated specific CTLs recognize, neutralize and destroy through cell lysis HER2 expressing cancer cells, including occult cancer cells and micrometastatic foci. The nelipepimut immune response can also generate CTLs to other immunogenic peptides through inter- and intra-antigenic epitope spreading. Based on a successful Phase 2 trial, which achieved its primary endpoint of DFS, the Food and Drug Administration (FDA) granted NeuVax a Special Protocol Assessment (SPA) for its Phase 3 PRESENT (Prevention of Recurrence in Early-Stage, Node-Positive Breast Cancer with Low to Intermediate HER2 Expression with NeuVax Treatment) study.

The active portion of the study will last three years (36 months). The follow-up will last from 5 to 10 years.

Endpoints:

1. Primary efficacy endpoint:

   * 3-year DFS
2. Secondary efficacy endpoints:

   * 5- and 10-year DFS
   * 3-year OS
   * 5- and 10-year OS
   * Safety profile, and adverse events (AEs)
   * Patterns of recurrence to include Time to recurrence (TTR), time to local recurrence (TTLR), time to distant recurrence (TTDR), time to bone metastases (TTBM)

Safety Assessments:

Subjects will be assessed at every study visit for the safety endpoints, AEs,vital signs, physical examinations and laboratory data; yearly follow-up of survival will include imaging studies, ECGs, MUGA or ECHO scans and concomitant medications.

ELIGIBILITY:
Key Inclusion Criteria:

* Pathological diagnosis of invasive adenocarcinoma of the breast
* Breast cancer completely excised, or patient receiving neoadjuvant therapy prior to surgery
* One of these 2 surgical treatments and axillary staging with sentinel lymph node dissection or axillary dissection level I/II:

  1. Total mastectomy-patients with a positive sentinel lymph node must have undergone a completion axillary dissection level I/II
  2. BCS (lumpectomy)-patients with a positive sentinel lymph node must have undergone a completion axillary dissection level I/II unless they had clinically node negative T1-T2 tumors and fewer than 3 involved lymph nodes
* Node-positive disease
* Primary tumor stage T1-3 at initial diagnosis
* HER2 negative (HER2 1+ by IHC or HER2 2+ by IHC/FISH)
* HLA-A2 or HLA-A3 haplotype
* Completed NCCN approved neo-adjuvant/adjuvant chemotherapy or both
* Completed radiation therapy
* No evidence of disease
* Able and willing (or have legal representative) to understand the study and provide consent

Key Exclusion Criteria:

* Bilateral breast malignancy or suspicious mass in opposite breast
* Inflammatory breast malignancy
* History of prior breast cancer, ductal carcinoma in situ
* Prior trastuzumab therapy
* New York Heart Association Stage 3 or 4 cardiac disease
* Sensory/motor neuropathy ≥ Grade 2
* Autoimmune diseases or immune deficiency disease
* Subjects on chronic steroid therapy, other immunosuppressive therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 758 (Actual)
Dates: Start 2011-11; Primary Completion 2016-09-21 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
Comparison of DFS in vaccine treated patients and control patients | 36 months
  The primary objective is to compare the DFS in subjects with operable early-stage, node-positive breast cancer who receive standard of care multimodality therapy plus NeuVax™ as the treatment group or standard of care multimodality therapy plus the vaccine adjuvant, Leukine® as the control group.

SECONDARY OUTCOMES:
Assessment of DFS and OS at 3, 5 and 10 years in vaccine and control groups, respectively; assessment of safety | 3 through 10 years
  The secondary objectives are to evaluate the 2 groups of subjects for:
  * 5- and 10-year DFS
  * 3-year OS
  * 5- and 10-year OS
  * Time to recurrence (TTR), time to local recurrence (TTLR), time to distant recurrence (TTDR), time to bone metastases (TTBM)
  * Overall safety profile and adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Mittendorf, MD,FACS, Principal Investigator — M.D. Anderson Cancer Center
Locations (197):
- United States (81):
  - Alabama Oncology, Bessemer, Alabama
  - Physicians Pain Specialists of Alabama, P.C., Mobile, Alabama
  - Pain Centers Nationwide, Peoria, Arizona
  - Valley Pain Consultants, Scottsdale, Arizona
  - East Valley Hematology and Oncology Medical Group, Burbank, California
  - Coastal Pain Research, Carlsbad, California
  - Navajo Road Pain Management Center, El Cajon, California
  - California Cancer Associates for Research and Excellence, Inc., Fresno, California
  - California Cancer Associates For Research and Excellence, Fresno, California
  - St. Jude Medical Center, Virginia K. Crosson Cancer Center, Fullerton, California
  - Interventional Pain Management, Irvine, California
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - University of Southern California/Norris Cancer Hospital, Los Angeles, California
  - Alexander Ford, MD, Los Angeles, California
  - Cancer Care Institute, Los Angeles, California
  - Pete J. Ruane, MD, Inc., Los Angeles, California
  - Cedars-Sinai Medical Center Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Moores UC San Diego Cancer Center (UCSD), San Diego, California
  - University of California, San Francisco (UCSF), Hellen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Pain Institute of Santa Monica, Santa Monica, California
  - Randy Scharlach, MD, Woodland Hills, California
  - University of Colorado Cancer Center, Anschutz Medical Campus, Aurora, Colorado
  - Red Rocks Center for Rehabilitation, Golden, Colorado
  - Western Connecticut Health Network, Danbury Hospital, Danbury, Connecticut
  - Stamford Hospital, Bennett Cancer Center, Stamford, Connecticut
  - Pain Management Associates of CT, PC, Stamford, Connecticut
  - Innovative Medical Research of South Florida, Inc., Aventura, Florida
  - Holy Cross Hospital-Michael & Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - Cancer Specialists of North Florida (ICON), Jacksonville, Florida
  - MD Anderson Center-Orlando Health, Orlando, Florida
  - Florida Cancer Research Institute (Florida Cancer Care), Plantation, Florida
  - Florida Cancer Care, Plantation, Florida
  - H.Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Interventional Spine and Pain Management, Atlanta, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Cancer Treatment Centers of America, Newnan, Georgia
  - Northwestern University Feinberg School of Medicine, Lynn Sage Comprehensive Breast Center, Chicago, Illinois
  - Pain Management Institute, Overland Park, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - James Graham Brown Cancer Center, University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Center of Cancer and Blood Disorders (VEEDA network), Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Department of Hematology and Oncology, Burlington, Massachusetts
  - Physiatry Consultants, Bay City, Michigan
  - Michigan Interventional Pain Center, Brownstown, Michigan
  - William Beaumont Hospital Cancer Center, Royal Oak, Michigan
  - Glenn Saperstein, D.O., LLC, Saginaw, Michigan
  - Advanced Physical Medicine, Saint Clair Shores, Michigan
  - Fountain Medical Group, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Upper East Side Pain Medicine, P.C., New York, New York
  - Comprehensive Pain Management, Syosset, New York
  - Eastchester Cancer Care Center, The Bronx, New York
  - APWI, Williamsville, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - St. Alexius Medical Center, Mid Dakota Clinic, PC, Bismarck, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Gettysburg Cancer Center, Hillsdale, Pennsylvania
  - Conemaugh Memorial Hospital-Memorial Medical Center, Johnstown, Pennsylvania
  - J. Fred Stoner, MD, New Castle, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Cancer Center, Pittsburgh, Pennsylvania
  - Progressive Pain Solutions, Wind Gap, Pennsylvania
  - Jerrold Rosenberg, MD, Providence, Rhode Island
  - The West Clinic Comprehensive Breast Center, Germantown, Tennessee
  - The West Clinic, Memphis, Tennessee
  - PRIDE, Dallas, Texas
  - UT Southwestern Medical Center / Simmons Comprehensive Cancer Center, Dallas, Texas
  - Brooke Army Medical Center (now SAMMC), Fort Sam Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Cancer Institute Research, Seattle, Washington
  - Multicare Health System-Research Institute, Tacoma, Washington
  - Medical College of Wisconsin Department of Surgery Froedtert Hospital and Cancer Center, Milwaukee, Wisconsin
- Bulgaria (5):
  - Central Onco Hospital, Plovdiv
  - Serdika, Sofia
  - Tsaritsa Yoanna - ISUL, Sofia
  - Sveta Marina, Varna
  - Complex Oncology Center, Veliko Tarnovo, Veliko Tarnovo
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Health Sciences North Cancer Centre, Greater Sudbury, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Hospital Charles LeMorne, Greenfield Park, Quebec
- Czechia (4):
  - Masaryk Memorial Cancer Institute, Comprehensive Cancer Care Clinic, Brno
  - University Hospital Hradec Kralove, Clinic of Oncology and Radiotherapy, Hradec Králové
  - University Hospital Olomouc, Clinic of Oncology, Olomouc
  - General University Hospital in Prague, Clinic of Oncology, Prague
- France (4):
  - Institut de Cancérologie de l'Ouest Siet Paul Papin, Angers, Cedex 9
  - Centre Oscar Lambret, Cédex, Lille
  - Institut de Cancérologie de l'Ouest/René Gauducheau, Saint Herblain, Nantes Cedex, Loire-Atlantique
  - Centre Antoine Lacassagne, Nice
- Germany (13):
  - Charité Campus Mitte Universitaetsmedizin-Berlin Brustzentrum/Studienzentrum, Berlin
  - Brustzentrum Klinikum Bremen-Mitte gGmbH, Bremen
  - Universitätsklinikum Erlangen, Frauenklinik, Erlangen
  - Kliniken Essen Mitte, Evang. Huyssens Stiftung/Knappschaft GmbH, Klinik für Senologie/Brustzentrum, Essen
  - Universitätsklinikum Frankfurt, Klinik für Frauenheilkunde und Geburtshilfe, Frankfurt
  - Nationales Centrum für Tumorerkrankungen (NCT), Gynäkologische Onkologie, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universität Marburg, Marburg
  - Rotkreuzklinikum München gGmbH, Frauenklinik, München
  - Universitätsklinikum Münster, Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Münster
  - Klinikum Stuttgart, Krankenhaus Bad Cannstatt, Frauenklinik, Stuttgart
  - Klinikum Mutterhaus der Borromaeerinnen, Trier
  - Gemeinschaftspraxis für Innere Medizin, Haematologie und internistische Onkologie Dr. R Schlag/Dr. Schoettker, Würzburg
- Hungary (6):
  - Hetenyi Geza Hospital, Department of Oncology, Szolnok, Jász-Nagykun-Szolnok
  - Szent Margit Hospital, V. Department of Internal Medicine, Oncology, Budapest
  - Semmelweis University, Department of Diagnostic Radiology and Oncotherapy, Budapest
  - Petz Aladar County Teaching Hospital, Center for Oncoradiology, Győr
  - Kaposi Mor County Teaching Hospital, Center for Clinical Oncology, Kaposvár
  - Borsod-Abauj-Zemplen County Hospital and University Educational Hospital, Center for Clinical Oncology and Radiology, Miskolc
- Israel (4):
  - Rambam Health Care Campus, Haifa, Haifa District
  - Sheba Medical Centre, Tel Hasomer, Ramat Gan
  - Rabin Medical Centre, Petah Tikva
  - Kaplan Medical Centre, Rehovot
- Poland (6):
  - Provincial Specialist Hospital in Wroclaw, Department of Chemotherapy, Kamienskiego, Wroclaw
  - Polish Red Cross Marine Hospital, Department of Chemotherapy, Gdynia
  - Nicolaus Copernicus Memorial Provincial Specialist Hospital in Lodz, Department of Chemotheraphy, Lodz
  - Greater Poland Cancer Center, Department of Chemotherapy, Poznan
  - Magodent, Warsaw
  - Non-Public Health Care Facility MAGODENT, Warsaw
- Romania (10):
  - "Gavril Curteanu" Municipal Clinical Hospital, Oradea, Bihor County
  - Medisprof SRL, Department of Medical Oncology, Cluj-Napoca, Cluj
  - Oncology Center "Sf. Nectarie", Department of Medical Oncology, Craiova, Dolj
  - Dr. Constantin Opris County Emergency Hospital, Department of Oncology, Baia Mare, Maramures
  - Filantropia Clinical Hospital, Obstetrics and Gynaecology Department, Bucharest
  - Coltea Clinical Hospital, Oncology Department, Bucharest
  - Bucharest Universtiy Emergency Hosptial, Oncology Department, Bucharest
  - "Prof. Dr. Ion Chiricuta" Institute of Oncology, Cluj-Napoca
  - Iasi Regional Oncology Institute, Department of Medical Oncology, Iași
  - Oncomed SRL, Department of Medical Oncology, Timișoara
- Russia (30):
  - Oncology Center #2, Department of Healthcare of Krasnodar Territory Administration, Sochi, Krasnodarskiy Kray
  - Republican Oncology Center, Saransk, Respublika Mordoviya
  - Pyatigorsk Oncology Center, Pyatigorsk, Stavropol Kray
  - Republican Clinical Oncoogy Center, Kazan', Tatarstan Republic
  - Arkhangelsk Clinical Oncology Center, Arkhangelsk
  - Regional Oncology Center, Irkutsk
  - Ivanovo Regional Oncology Center, Ivanovo
  - Clinical Oncology Center #1, Department of Healthcare of Krasnodar Territory Administration, Krasnodar
  - Krasnoyarsk Kryzhanovsky Regional Oncology Center, Krasnoyarsk
  - Kursk Regional Clinical Oncology Center, Kursk
  - N.N. Blokhin Russian Cancer Research Center, Moscow
  - N.N. Blokhin Russian Cancer Reserach Center, Moscow
  - Clinical Diagnostics Center, Nizhny Novgorod
  - Nizhny Novgorod Regional Oncology Center, Nizhny Novgorod
  - Orenburg Regional Clinical Oncology Center, Orenburg
  - Orel Oncology Center, Oryol
  - Medical Institution of Ryazan Region, Ryazan
  - Leningrad Regional Oncology Center, Saint Petersburg
  - St. Petersburg Clinical Hospital, Saint Petersburg
  - Mechnikov North-Western State Medical University, Saint Petersburg
  - Petrov Research Institute of Oncology, Saint Petersburg
  - Municipal Clinical Oncology Center, Saint Petersburg
  - Samara Regional Clinical Oncology Center, Samara
  - Tambov Regional Clinical Oncology Center, Tambov
  - Research Institute of Oncology, Tomsk
  - Bashkir State Medical University, Ufa
  - Regional Clinical Oncology Center, Veliky Novgorod
  - Volgograd Regional Oncology Center #3, Volzhskiy
  - Yaroslavl Regional Oncology Center, Yaroslavl
  - Sverdlovsk Regional Oncology Center, Yekaterinburg
- Ukraine (17):
  - Clinical Diagnostics Center, Simferopol, Autonomous Republic of Crimea
  - Kryvyi Rih Oncology Center/Dnipropetrovsk Regional Council, Department of Chemotherapy, Kryvyi Rih, Dnipropetrovsk Oblast
  - Mariupol City Interdistrict Oncology Center, Surgery Department #2, Mariupol, Donetsk Oblast
  - Kharkiv Regional Clinical Oncology Center, Day Care Unit, Kharkiv, Kyivskyi District
  - Chernivtsi Regional Clinical Oncology Center, Day Care Unit, Chernivtsi
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4/Dnipropetrovsk Regional Council, Department of Chemotherapy, Dnipropetrovsk
  - Donetsk City Oncology Center, Donetsk
  - Donetsk Regional Antitumor Center, Oncosurgery Department #2, Donetsk
  - State Institution: S.P. Grigoriev Institute of Medical Radiology Under the Academy of Medical Sciences of Ukraine, Kharkiv
  - Public Institution: Kiev Regional Oncology Hospital within Kyiv Regional Council, Kiev
  - Kirovohrad Regional Oncology Center, Department of Mammology, Kirovohrad
  - Kyiv City Clinical Oncology Center, Department of Chemotherapy, Kyiv
  - Lviv State Regional Treatment and Diagnostics Oncology Center, Department of Chemotherapy, Lviv
  - Odesa Regional Clinical Hospital, Center for Mastology, Odesa
  - Zakarpattia Regional Clinical Oncology Center, Department of Chemotherapy, Uzhhorod
  - Vinnytsia Regional Clinical Oncology Center, Vinnytsia
  - Public Institution Zaporizhia Regional Clinical Oncology Center within Zaporizhia Regional Council, Zaporizhia
- United Kingdom (12):
  - Macclesfield District General Hospital, Macclesfield, Cheshire
  - The Christie NHS Foundation Trust, Withington, Manchester
  - James Cook University Hospital, Middlesbrough, Middlesborough
  - Plymouth Oncology Centre, Derriford Hospital, Plymouth, Plymouth
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Leeds Teaching Hospitals Trust, St. James University Hospital, Leeds, West Yorkshire
  - Leicester Royal Infirmary, Leicester
  - The Royal Marsden NHS Foundation Trust, London
  - Academic Unit of Oncology, Nottingham University Hospital-City Campus, Nottingham
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - University Hospital of North Staffordshire, Stoke-on-Trent

REFERENCES:
- [Background] Amin A, Benavides LC, Holmes JP, Gates JD, Carmichael MG, Hueman MT, Mittendorf EA, Storrer CE, Jama YH, Craig D, Stojadinovic A, Ponniah S, Peoples GE. Assessment of immunologic response and recurrence patterns among patients with clinical recurrence after vaccination with a preventive HER2/neu peptide vaccine: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer Immunol Immunother. 2008 Dec;57(12):1817-25. doi: 10.1007/s00262-008-0509-2. Epub 2008 Apr 8. PMID 18392824
- [Background] Mittendorf EA, Clifton GT, Holmes JP, Clive KS, Patil R, Benavides LC, Gates JD, Sears AK, Stojadinovic A, Ponniah S, Peoples GE. Clinical trial results of the HER-2/neu (E75) vaccine to prevent breast cancer recurrence in high-risk patients: from US Military Cancer Institute Clinical Trials Group Study I-01 and I-02. Cancer. 2012 May 15;118(10):2594-602. doi: 10.1002/cncr.26574. Epub 2011 Oct 11. PMID 21989902
- [Derived] Mittendorf EA, Lu B, Melisko M, Price Hiller J, Bondarenko I, Brunt AM, Sergii G, Petrakova K, Peoples GE. Efficacy and Safety Analysis of Nelipepimut-S Vaccine to Prevent Breast Cancer Recurrence: A Randomized, Multicenter, Phase III Clinical Trial. Clin Cancer Res. 2019 Jul 15;25(14):4248-4254. doi: 10.1158/1078-0432.CCR-18-2867. Epub 2019 Apr 29. PMID 31036542
- See also: Sponsor website — http://www.galenabiopharma.com
- See also: Vaccine site — http://NeuVax.com